CLINICAL TRIAL: NCT04500444
Title: Effects of Blood Flow Restricted Aerobic Exercise on Pain, Functional Status, Quality of Life, and Hormonal Response to Exercise in Fibromyalgia Patients - Randomized Controlled Trial
Brief Title: Effects of Aerobic Exercise Training With and Without Blood Flow Restriction in Fibromyalgia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Mert Zure, Medical Doctor, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1301
Record Dates: First submitted 2020-08-03; First posted 2020-08-05 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Fibromyalgia
Keywords: blood flow restriction training; fibromyalgia; aerobic training
MeSH Terms: conditions — Fibromyalgia | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blood-Flow Restriction Group (Experimental): An aerobic exercise program with blood flow restriction will be applied 4 times a week for a total of 6 weeks. The aerobic exercise training consists of a warm up period for 5 minutes, walking on treadmill at 4 km per hour speed for 20 minutes and cooling down for another 5 minutes. The blood flow restriction protocol will be applied to both lower extremities at the crotch level with 10 cm wide elastic bandages before warming up. Before the first application, patients will be evaluated by a specialist physician using ultrasonography and it will be ensured that the arterial blood flow is not restricted as the blood flow restriction restricts only venous blood flow. The pressure threshold at this point is the level to be used in subsequent training sessions and the same person (physician) will be bandaging in the same way during all subsequent training sessions.
  Interventions: Other: exercise training
- Control Group (Sham Comparator): An aerobic exercise program with blood flow restriction will be applied 4 times a week for a total of 6 weeks. The aerobic exercise training consists of a warm up period for 5 minutes, walking on treadmill at 4 km per hour speed for 20 minutes and cooling down for another 5 minutes. The sham blood flow restriction protocol will be applied which consists of loose bandaging to both lower extremities at the crotch level with 10 cm wide elastic bandages before warming up. The same person (physician) will be bandaging in the same way during all subsequent training sessions. The pressure feeling of the patient must correspond to level 0 -not tight at all- before starting the exercise training.
  Interventions: Other: exercise training

INTERVENTIONS:
Other: exercise training — An aerobic exercise program with blood flow restriction will be applied 4 times a week for a total of 6 weeks. The aerobic exercise training consists of a warm up period for 5 minutes, walking on treadmill at 4 km per hour speed for 20 minutes and cooling down for another 5 minutes.
  Other Names: low intensity aerobic training

SUMMARY:
In our study, we aimed to evaluate and compare the effects of low-intensity aerobic exercise training with blood flow restriction and without blood flow restriction, on pain, functional status, quality of life and catecholamine metabolite levels in 24-hour urine in adults with Fibromyalgia.

DETAILED DESCRIPTION:
Fibromyalgia is a chronic disorder characterized by widespread pain, fatigue, sleep disturbance, cognitive disorder and other physical symptoms that negatively affect physical and sensory functions and impair quality of life. [1]

Fibromyalgia is seen in the society at 2-4%, and the ratio of women to men is 9:1. It is seen most often between the ages of 45 and 60. Neuroendocrine deviations arise with the contribution of central sensitization and / or peripheral pain mechanisms as a result of environmentally related physiological and psychological stresses of people with genetic predisposition.[2]

The depletion of biogenic amines in the central nervous system is blamed on the basis of major symptoms such as musculoskeletal pain, muscle fatigue, sleep disturbance, and comorbid chronic depression, anxiety, migraine, which are clinically observed in fibromyalgia. Decreased levels of aminergic neurotransmitters is detected in cerebrospinal fluid (CSF) of fibromyalgia patients, especially serotonin, dopamine, norepinephrine.[3]

Studies have found that different exercise programs have positive effects on pain and functionality in fibromyalgia cases, and no side effects of these exercise programs have been observed. Aerobic exercise training is one of the most studied exercise modalities in fibromyalgia patients.[4]

However, an increase in post-exercise pain was also found in patients with fibromyalgia due to a decrease in muscle blood flow, defect in muscle contraction physiology and a change in post-exercise pain modulation. In addition, it has been reported that the hormone response given to the exercise is impaired. All of these disorders can decrease patients' compliance to exercise.[5]

Exercise with blood flow restriction - Blood Flow Restriction Training (BFRT) - is an increasingly popular exercise modality that creates a physiological effect equivalent to a high exercise intensity when exercising at low exercise intensities. In current studies, although a similar response to high-intensity aerobic exercise was obtained by performing low-intensity blood flow-restricted aerobic exercise training in other patient groups, a recommendation regarding the use of BFRT in a specific disease such as fibromyalgia is lacking.[6]

In our study, we aimed to evaluate and compare the effects of low-intensity aerobic exercise training with blood flow restriction and without blood flow restriction, on pain, functional status, quality of life and catecholamine and melatonin metabolite levels in 24-hour urine in adults with Fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

1. Being between 18 and 55 years old
2. Symptoms lasting longer than 3 months
3. According to the 2016 ACR criteria, the Common Pain Scale Score is ≥7 and the Symptom Severity Score is ≥5 or according to the 2016 ACR criteria, the Symptom Severity Score is ≥9 and the Common Pain Scale Score is between 4-6.
4. Fibromyalgia Impact Questionnaire (FIQ) score between 35 and 65 (out of 100)
5. To be able to come to the hospital for treatment 4 days a week for 6 weeks.
6. No change in the medical treatment received due to fibromyalgia syndrome during the study

Exclusion Criteria:

1. Presence of known central nervous system or peripheral nervous system disease, progressive neurological deficit
2. Peripheral venous insufficiency and coagulopathies
3. Serious cardiovascular pathologies
4. Sensory loss, loss of position sensation, unhealed fracture or open surgical wound
5. Uncontrolled hypertension, diabetes
6. Cognitive disorder causing simple commands difficulty
7. Pregnancy
8. Having entered the menopause

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-11-13 (Actual); Primary Completion 2020-09-18 (Estimated); Study Completion 2020-12-18 (Estimated)

PRIMARY OUTCOMES:
Change in Fibromyalgia Impact Questionnaire (FIQ) score | Baseline, Immediately after the intervention , 3 months after the intervention period
  The Fibromyalgia Impact Questionnaire (FIQ) was developed by clinicians at the Oregon Health Sciences University in the late 1980s to capture and evaluate the total spectrum of fibromyalgia-related problems and response to treatment. It was first used in 1991 and is still an indicator of therapeutic effectiveness today. it is used frequently.
  It consists of 10 questions to measure physical, emotional, cognitive and motivational symptoms such as physical disability, pain, fatigue, joint stiffness, depression and anxiety in fibromyalgia. Each question has been scored within itself.
  The total score will be between 0-100. 100 points indicate the highest exposure to the disease.

SECONDARY OUTCOMES:
Change in Central Sensitization Inventory Score | Baseline, Immediately after the intervention , 3 months after the intervention period
  Central Sensitization Inventory (CSI) is a scale used to detect patients with symptoms associated with central sensitization or types of central sensitization syndrome such as fibromyalgia, temporomandibular joint disease, tension type headache, migraine.
  The Central Sensitization Inventory (CSI) consists of two parts:
  Part A consists of 25 questions about central sensitization syndrome (CNS) symptoms; Section B examines the patient's condition of being diagnosed with certain CNS diseases or CNS related diseases such as anxiety and depression.
  The patient answers 25 questions in section A with a score between 0 and 4. The total score will be between 0-100. Results above 40 points indicate central sensitization.
Change in Visual Analog Scale for Pain | Baseline, Immediately after the intervention , 3 months after the intervention period
  This scale is used to assess pain subjectively. Scale consists of a 10 cm long horizontal line. The two ends are named differently. 0 means no pain, 10 means the most severe pain.
  The patient is asked to mark a point on this line that corresponds to the severity of pain he feels. The distance between the marked point and the lowest end of the line is measured and the numerical value found shows the pain intensity of the patient.
Change in Beck Depression Inventory Score | Baseline, Immediately after the intervention , 3 months after the intervention period
  Beck Depression Criterion (BDI) is a commonly used evaluation criterion for diagnosis and follow-up parameters in assessing depression status.
  It contains 21 categories to measure physical, emotional, cognitive and motivational symptoms such as hopelessness, irritability, guilt, feeling of punishment, fatigue, and weight loss in each depression, and each category is scored between 0-3. The patient is asked to mark the most appropriate one for the four options in each category. Scoring progressively increases from the absence of symptoms to severe symptoms. 0-10 points: No depression, 11-17 points: Mild depression, 18-23 points: Moderate depression, 24 and above points: Severe depression.
Change in Chronic Pain Acceptance Questionnaire - 8 Score | Baseline, Immediately after the intervention , 3 months after the intervention period
  CPAQ-8 is an 8-question survey. It measures the level of patient acceptance of pain and the level of continuing social, daily activities. Each question is scored between 0-5. The higher the score, the higher the pain acceptance level.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşegül Ketenci, Principal Investigator — Professor
Locations (1):
- Istanbul University Istanbul Faculty of Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Evcik D, Ketenci A, Sindel D. The Turkish Society of Physical Medicine and Rehabilitation (TSPMR) guideline recommendations for the management of fibromyalgia syndrome. Turk J Phys Med Rehabil. 2019 May 28;65(2):111-123. doi: 10.5606/tftrd.2019.4815. eCollection 2019 Jun. PMID 31453551
- [Background] Hauser W, Ablin J, Fitzcharles MA, Littlejohn G, Luciano JV, Usui C, Walitt B. Fibromyalgia. Nat Rev Dis Primers. 2015 Aug 13;1:15022. doi: 10.1038/nrdp.2015.22. PMID 27189527
- [Background] Singh L, Kaur A, Bhatti MS, Bhatti R. Possible Molecular Mediators Involved and Mechanistic Insight into Fibromyalgia and Associated Co-morbidities. Neurochem Res. 2019 Jul;44(7):1517-1532. doi: 10.1007/s11064-019-02805-5. Epub 2019 Apr 19. PMID 31004261
- [Background] Michiels V, Cluydts R. Neuropsychological functioning in chronic fatigue syndrome: a review. Acta Psychiatr Scand. 2001 Feb;103(2):84-93. doi: 10.1034/j.1600-0447.2001.00017.x. PMID 11167310
- [Background] Bidonde J, Busch AJ, Bath B, Milosavljevic S. Exercise for adults with fibromyalgia: an umbrella systematic review with synthesis of best evidence. Curr Rheumatol Rev. 2014;10(1):45-79. doi: 10.2174/1573403x10666140914155304. PMID 25229499
- [Background] Genc A, Tur BS, Aytur YK, Oztuna D, Erdogan MF. Does aerobic exercise affect the hypothalamic-pituitary-adrenal hormonal response in patients with fibromyalgia syndrome? J Phys Ther Sci. 2015 Jul;27(7):2225-31. doi: 10.1589/jpts.27.2225. Epub 2015 Jul 22. PMID 26311959
- [Background] Patterson SD, Hughes L, Head P, Warmington S, Brandner C. Blood flow restriction training: a novel approach to augment clinical rehabilitation: how to do it. Br J Sports Med. 2017 Dec;51(23):1648-1649. doi: 10.1136/bjsports-2017-097738. Epub 2017 Jun 22. No abstract available. PMID 28642225